CLINICAL TRIAL: NCT04375410
Title: Re-opening of the Country and Dermal Consequences of Mandatory Intensified Handwash and Hand Disinfection Among a Danish Pediatric Population During the COVID19 Pandemic
Brief Title: Consequences of Intensified Handwash and Hand Disinfection Among Children During the COVID19 Pandemic
Status: Completed | Type: Observational
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Tine Caroc Warner, Principal investigator, Regionshospital Nordjylland
Other Study IDs: SH042020
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hand Eczema; Hand Dermatitis; Covid19
Keywords: Dermatitis; Hand wash; Hand disinfection; Children; Pediatric
MeSH Terms: conditions — COVID-19; Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID-19 pandemic after reopening of the country, school, kindergarten and daycare, children have been obligated to do frequent handwash. The study group wished to investigate whether this has had implications on symptoms of dry, red, itchy or sore hands and hand eczema. The investigation was performed within the first and second week after reopening by questionnaires distributed to parents electronically via schools, kindergartens and daycare facilities electronic platforms.

DETAILED DESCRIPTION:
During the COVID-19 pandemic Denmark closed down, including schools, kindergartens and daycare. After reopening of the country 5 weeks later obligatory frequent handwash was a requirement from the government and routines has been implemented at all reopened schools, kindergartens and daycare. The study group wished to investigate whether this has had implications on symptoms of dry, red, itchy or sore hands and hand eczema. Also the study group wished to investigate if frequency or use of hand disinfection mattered. The investigation was performed within the first and second week after reopening by questionnaires distributed to parents electronically via schools, kindergartens and daycare electronic platforms. The questionnaire included 20 questions on demographics, frequency of hand wash and use of disinfectants, current and previous symptoms of eczema, atopic dermatitis and dispositions.

ELIGIBILITY:
Inclusion Criteria:

* All children returned to daycare, kindergarten or school after covid19 close down of the country

Exclusion Criteria:

* None

Ages: 0 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: Children i Hjoerring, Aalborg, Rebild or Skanderborg municipaility
Sampling Method: Non-Probability Sample
Enrollment: 6273 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Dermal reaction to frequent hand wash and disinfection in children | 9 days
  Dermal symptoms as a result of frequent hand wash and disinfection among children

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Haghstroem, M.D, PhD, Principal Investigator — Aalborg University Hospital, Aalborg University; Luise Borch, M.D, PhD, Principal Investigator — Regional Hospital West Jutland, Herning
Locations (1):
- Tine Caroc Warner, Hjørring, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borch L, Thorsteinsson K, Warner TC, Mikkelsen CS, Bjerring P, Lundbye-Christensen S, Arvesen K, Hagstroem S. COVID-19 reopening causes high risk of irritant contact dermatitis in children. Dan Med J. 2020 Aug 6;67(9):A05200357. PMID 32800064